CLINICAL TRIAL: NCT04780295
Title: COvid-19 REgistry on THROMBOSIS Complications Associated With Hospitalization
Brief Title: Coronavirus Disease (COvid-)19 REgistry on THROMBOSIS Complications
Acronym: CORE-THROMB
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Stavros Konstantinides, MD, Prof Stavros Konstantinides, MD, Medical Director of the, Johannes Gutenberg University Mainz
Other Study IDs: CTH C010; DRKS00022277 (Registry Identifier: DRKS (Deutsches Register klinischer Studien, engl.: German Clinical Studies Register))
Record Dates: First submitted 2021-02-09; First posted 2021-03-03 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: Covid19; thromboembolism; thromboprophylaxis; pulmonary embolism; anticoagulation
MeSH Terms: conditions — COVID-19; Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This online-based, observational retrospective registry aims to (i) study the rate of cardiovascular events, encompassing venous thromboembolic and arterial events, in consecutive hospitalized patients with coronavirus (Covid19), (ii) investigate the prevalent use of thromboprophylaxis, (iii) describe the use of imaging tests for the detection of cardiovascular events in patients with Covid19. This will also facilitate and constitute the basis for the conduction of interventional thromboprophylaxis studies in patients with Covid19.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients aged ≥ 18 years with a positive test for severe acute respiratory syndrome corona virus 2 (SARS-CoV2)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given the observational nature of this registry, no exclusion criteria will be applied.
Sampling Method: Probability Sample
Enrollment: 2708 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Fatal or non-fatal venous thromboembolism (VTE) | during index hospitalization for Covid19
  Rate of thromboembolic events encompassing pulmonary embolism (PE) and deep vein thrombosis (DVT)
Fatal or non-fatal cardiovascular events | during index hospitalization for Covid19
  Rate of cardiovascular events encompassing stroke and myocardial infarction
All-cause death | during index hospitalization for Covid19
  Rate of death from any cause

SECONDARY OUTCOMES:
Prevalence of cardiovascular risk factors | at baseline/enrollment
  Baseline prevalence of cardiovascular risk factors and use of specific medications (statins, Angiotensin-converting enzyme [ACE] inhibitors)
Length of hospitalization | first index hospitalization for Covid19
  Duration of inpatient stay
Prevalent use of in-hospital thromboprophylaxis | during index hospitalization for Covid19
  Use of unfractionated heparin (UFH), low-molecular weight heparin (LMWH), or direct oral anticoagulants (DOAC) on/after admission due to Covid19
In-hospital course of D-dimer (μg/mL) | during index hospitalization for Covid19
  Course of laboratory biomarker
In-hospital course of Troponin (ng/ml) | during index hospitalization for Covid19
  Course of laboratory biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Konstantinides, MD, Prof, Study Chair — University Medical Center Mainz, Johannes Gutenberg University Mainz
Locations (30):
- Brazil (3):
  - Unicamp (Universidade Estadual de Campinas; University of Campinas), Campinas
  - Hospital Sírio-Libanês, São Paulo
  - Hospital de Campanha Anhembi, São Paulo
- Amager and Hvidovre Hospital, Hvidovre, Denmark
- Germany (9):
  - Universitätsklinikum Koeln, Cologne
  - Augusta-Krankenhaus Duesseldorf, Düsseldorf
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum des Saarlandes und Medizinische Fakultät der Universität des Saarlandes, Homburg
  - DRK Kliniken Berlin Köpenick, Köpenick
  - Universitätsmedizin Mainz, Mainz
  - Krankenhaus Neuwittelsbach, Munich
  - Paracelsus Medizinische Privatuniversität am Klinikum Nuernberg, Nuremberg
  - DRK Kliniken Berlin Westend, Westend
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (13):
  - University of Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale (ASST) Lariana, Como
  - Ospedale Sacra Famiglia Fatebenefratelli, Erba
  - Presidio Ospedaliero Santa Croce di Fano, Fano
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Civile di Guastalla - Azienda Unità Sanitaria Locale (AUSL) Reggio Emilia, Guastalla
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Maggiore di Parma - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Civile di Castel San Giovanni - Azienda Unità Sanitaria Locale (AUSL) di Piacenza, Piacenza
  - Santa Maria Nuova Hospital - Azienda Unità Sanitaria Locale (AUSL) IRCCS di Reggio Emilia, Reggio Emilia
  - IRCCS Humanitas Clinical and Research Hospital, Rozzano
  - Università degli studi dell' Insubria (University of Insubria), Varese
- Instituto Nacional de Cardiologia Ignacio Chavez (National Institute of Cardiology Igancio Chavez), Mexico City, Mexico
- Hospital Quirónsalud, Málaga, Spain
- Erdem Medical Center, Istanbul, Turkey (Türkiye)